CLINICAL TRIAL: NCT06359899
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Study to Investigate the Efficacy, Safety and Tolerability of Oral Administered AK0901 Capsules in Children Aged 6-12 Years Old With Attention Deficit Hyperactivity Disorder
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of Oral AK0901 in Children With ADHD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK0901-2001
Record Dates: First submitted 2024-03-25; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — serdexmethylphenidate and dexmethylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AK0901 cohort (Experimental): 13.1 mg/2.6 mg AK0901, 26.1 mg/5.2 mg AK0901, 39.2 mg/7.8 mg AK0901
  Interventions: Drug: AK0901 capsule
- Placebo cohort (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK0901 capsule — Active Substance: AK0901, Pharmaceutical Form: Capsule, Route of Administration: Oral
  Other Names: AZSTARYS (SDX/d-MPH capsules)
  Arms: AK0901 cohort
Drug: Placebo — Active Substance: Placebo, Pharmaceutical Form: Capsule, Route of Administration: Oral
  Arms: Placebo cohort

SUMMARY:
This study is a Phase 3, multicenter, dose-optimized, double-blind, randomized, placebo-controlled study designed to evaluate the efficacy, safety, and tolerability of oral AK0901 capsules in children 6 to 12 years old with Attention Deficit Hyperactivity Disorder（ADHD）.

DETAILED DESCRIPTION:
The study consists of an approximately 28-day screening period, a 28-day double-blind treatment period, and a follow-up period for 5±2 days.

During the screening period, all subjects must sign an informed consent form and complete all assessment items at the screening visit prior to the screening. Study drug is started within 28 days of signing the informed consent form.

During the double-blind treatment period, all eligible subjects are randomized 1:1 to receive AK0901 or placebo once daily for 4 weeks. During the first week, all subjects are given a starting dose of 39.2 mg/7.8 mg AK0901 or matching placebo; from the second week, the dose drug can be increased or decreased, or maintained at the original dose level at weekly follow-up depending on tolerability and optimal individual dose response at the investigator's discretion.

After the last dose in the double-blind treatment period, subjects will enter a 5 ± 2 day follow-up period for safety assessments. The primary analysis will be performed after all subjects have completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing informed consent form, subjects must be between 6 and 12 years of age (inclusive) and of any gender.
2. Subjects meet the diagnostic criteria for ADHD (attention deficit or hyperactivityj/impulsivity or combined attention deficit and hyperactivity/impulsivity manifestations) in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) as medically evaluated and confirmed by the Chinese version of Kiddie-schedule for affective disorders and schizophrenia-present and lifetime version DSM-5 (K-SADS-PL-C DSM-5).
3. An ADHD-RS-5 total score of at least 28. For subjects requiring washout of ADHD medications, this criterion refers to a score following washout.
4. A score of at least 3 (mildly ill) on the Clinical Global Impressions - Severity (CGI-S) scale as assessed by clinician. For subjects requiring washout of ADHD medications, this criterion refers to a score following washout.
5. Weight exceeds the median weight for the appropriate age and sex minus two times the standard deviation (2SD) .
6. Able to sign the ICF, including compliance with the requirements and limitations specified in the ICF and this protocol.
7. Understand the importance of adhering to study medication requirements and completing all assessments on time throughout the study, and agree to strictly follow the requirements as specified in the protocol, including restrictions on concomitant medications during the study.
8. The subject's parent/legal guardian must ensure that the subject: has washed out ongoing stimulants for ADHD and herbal/Chinese patent medicines for the treatment of ADHD 5 days prior to the first dose and is abstained from these medications until the end of the study or early termination of the study; and must wash out ongoing non-stimulants for ADHD 14 days prior to the first dose and is abstained from these medications until the end of the study or early termination of the study.

Exclusion Criteria:

Medical disorders

1. Pre-existing or current clinically significant disease or any condition that, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of study results, or would result in the subject's inability to complete study in accordance with the protocol.
2. Presence of evidence of central nervous system (CNS) diseases (e.g., tumor, inflammation, epilepsy, vascular disease), or neuromuscular disorder that may have occurred in childhood (e.g., Duchenne muscular dystrophy, myasthenia gravis), or history of persistent neurological symptoms that can be attributed to severe head injury, or other serious nervous system disorders. Simple febrile seizure is allowed. Patients with electroencephalogram suggesting epileptiform discharge or seizure susceptibility will be excluded.
3. History of mental illness including, but not limited to, a diagnosis of bipolar disorder, major depressive disorder, conduct disorder, obsessive-compulsive disorder, childhood schizophrenia, autism spectrum disorder, disruptive mood dysregulation disorder (DMDD), intellectual developmental disorder, tic disorders, generalized anxiety disorder or panic disorder, severe sleep disorder, and genetic disorders associated with cognitive and/or behavioral disorder. Oppositional defiant disorder (ODD) is permitted if the condition is mild-moderate, not a current treatment priority, and the investigator assesses that the subject is appropriate and cooperative.
4. Subject has any history of attempted suicide or clinically significant suicidal ideation based on the Columbia-Suicide Severity Rating Scale (C-SSRS) assessment, in the opinion of the investigator, at screening or Day 1.
5. Cardiovascular system , digestive system , endocrine system, ophthalmology , respiratory system, and hepatic or renal system, or any other clinically significant concomitant diseases that could jeopardize the safety of the subject or affect the results of the study.
6. Active malignancy and/or history of malignancy.
7. History of allergy or suspected allergy to methylphenidate, serdexmethylphenidate, or AK0901 excipients.
8. History of serious allergy to any drug, or known history of allergy to more than one drug.

   Previous therapies/concomitant treatment
9. Have received or are receiving systematic cognitive behavioral therapy (CBT), behavioral therapy, or other non-drug therapies for ADHD within 1 month prior to screening.
10. Subject has taken ADHD medications from more than one class within 30 days prior to screening. Subjects on a stable dose of one ADHD medication with occasional use of ADHD medications from another class are exceptional at the discretion of the investigator.
11. Subjects with lack of response or intolerability to previous adequate dose and duration of treatment with methylphenidate products in the opinion of the investigator.
12. Use of monoamine oxidase inhibitors within 14 days prior to the first dose; use of the following medications within 21 days prior to the first dose: antidepressants, mood stabilizers, antipsychotics, coumarin anticoagulants, anticonvulsants, halogenated anesthetics, phenylbutazone, and sedative hypnotics.
13. Planned use of prohibited drugs or non-drug therapies as specified in the protocol during the study.

    Clinical study experience of prior/concomitant medications
14. Subject has participated in clinical study of any other investigational product within 90 days or 5 half-lives, whichever is longer, prior to screening, or is currently participating in another drug clinical trial.

    Diagnostic assessments
15. At the discretion of the investigator, has a clinically significant abnormal finding in the physical examination, neurological examination, vital signs, ECG, or clinical laboratory tests at screening.
16. Mean systolic or diastolic blood pressure measurements ≥ 95th percentile for corresponding age, gender, and height at screening or Day 1.
17. Electrocardiogram shows QTcF interval ≥ 450 ms at screening [QTcF = QT/(RR^0.33)].
18. Glutamic-pyruvate transaminase (SGPT) or glutamic-oxaloacetic transferase (SGOT) ≥ 1.5 × the upper limit of normal (ULN) or blood creatinine > ULN at screening.
19. Thyroid stimulating hormone (TSH), free thyroxine (FT4), or free tri-iodothyronine (FT3) abnormality at screening.

    Other exclusion criteria
20. Subjects with a history of drug or alcohol abuse within 1 year prior to screening; positive alcohol or drug screen at screening or Day 1 ;
21. Positive screening for methylphenidate at screening or Day 1.
22. Use of tobacco or other nicotine-containing products at screening.
23. Family history (parents and siblings) of sudden cardiac death, severe ventricular arrhythmia, or QT prolongation.
24. The subject's parent/legal guardian is an investigator of this study, employee of the study site with direct involvement in this study or any other studies under the direction of the investigator, sponsor's employee, or any family members of the investigator of this study, employee of study site or sponsor's employee.
25. Subject and parent/legal guardian are unable to communicate well with the investigator.
26. Any other reason that, in the opinion of the investigator, would make subject's participation inappropriate.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of AK0901 compared to placebo in children 6 to 12 years old with ADHD. | From Baseline (Pre-dose on Day 1) to week 3
  Change from baseline in ADHD-RS-5* total score at Week 3. Attention-Deficit Hyperactivity Disorder Rating Scale 5 is a scale containing 18 symptomatic entries with each entry scored on a 4-point scale. Each entry is scored using a frequency assessment from 0 (symptom never or rarely) to 3 (symptom very frequent), with a total score ranging from 0 to 54.
  A decreasing value of the total score represents a clinical improvement. Unless otherwise noted, the last non-missing measurement/assessment before the first dose of the investigational product is defined as the Baseline measurement. If a measurement/evaluation is performed on the same day of the first dose of the investigational product, these measurements will be considered as Baselines.

SECONDARY OUTCOMES:
Change from baseline in ADHD-RS-5 total score at Week 4. | From Baseline (Pre-dose on Day 1) to week 4
  Attention-Deficit Hyperactivity Disorder Rating Scale 5 is a scale containing 18 symptomatic entries with each entry scored on a 4-point scale. Each entry is scored using a frequency assessment from 0 (symptom never or rarely) to 3 (symptom very frequent), with a total score ranging from 0 to 54.
  A decreasing value of the total score represents a clinical improvement. Unless otherwise noted, the last non-missing measurement/assessment before the first dose of the investigational product is defined as the Baseline measurement. If a measurement/evaluation is performed on the same day of the first dose of the investigational product, these measurements will be considered as Baselines.
Changes in ADHD-RS-5 inattention subscale score from baseline to each visit in the Double-Blind Treatment Period | From Baseline (Pre-dose on Day 1) to week 4
  Attention-Deficit Hyperactivity Disorder Rating Scale 5 is a scale containing 18 symptomatic entries with each entry scored on a 4-point scale. Each entry is scored using a frequency assessment from 0 (symptom never or rarely) to 3 (symptom very frequent), with a total score ranging from 0 to 54.The 18 entries in the ADHD-RS-5 can be divided into two 9-item subscales, one to assess impulsivity-hyperactivity and the other to assess attention deficits.A decreasing value of the total score represents a clinical improvement.
Changes in ADHD-RS-5 hyperactivity/impulsivity subscale score from baseline to each visit in the Double-Blind Treatment Period. | From Baseline (Pre-dose on Day 1) to week 4
  Attention-Deficit Hyperactivity Disorder Rating Scale 5 is a scale containing 18 symptomatic entries with each entry scored on a 4-point scale. Each entry is scored using a frequency assessment from 0 (symptom never or rarely) to 3 (symptom very frequent), with a total score ranging from 0 to 54.The 18 entries in the ADHD-RS-5 can be divided into two 9-item subscales, one to assess impulsivity-hyperactivity and the other to assess attention deficits.A decreasing value of the total score represents a clinical improvement.
Change in CGI-S score from baseline to each visit in the Double-Blind Treatment Period | From Baseline (Pre-dose on Day 1) to week 4
  Clinical Global Impressions - Severity is a clinical rating scale used to assess the severity of psychopathology (ADHD symptoms in this study) on a scale from 1 to 7.A decreasing value of the score represents a clinical improvement.
CGI-I scores from V3 at each visit in the Double-Blind Treatment Period | From V3 (week 1) to week 4
  Clinical Global Impressions - Improvement is a clinical rating scale used to assess the degree of improvement in psychopathology (ADHD symptoms in this study) on a scale from 1 to 7. A decreasing value of the score represents a clinical improvement.
Change in WREMB-R score from baseline to each visit in the Double-Blind Treatment | From Baseline to week 4
  Weekly Rating of Evening and Morning Behavior - Revised is an 11-entry questionnaire to assess behavioral severity in the morning (3 entries) and evening (8 entries). Scores for each entry range from 0 to 3. A decreasing value of the total score represents a clinical improvement.
Proportion of subjects with adverse events (AEs) occurring during the study | From Baseline to Day 33
  To evaluate the safety and tolerability of AK0901.
Proportion of subjects with serious adverse events (SAEs) occurring during the study | From Baseline to Day 33
  To evaluate the safety and tolerability of AK0901.
Changes in respiratory rate during the study | From Baseline to Day 33
  To explore the difference in respiratory rate (bpm) with clinical significance between subjects on AK0901 and those on placebo.
Changes in heart rate during the study | From Baseline to Day 33
  To explore the difference in heart rate/pulse (bpm) with clinical significance between subjects on AK0901 and those on placebo.
Changes in body temperature during the study | From Baseline to Day 33
  To explore the difference in body temperature (Celsius) with clinical significance between subjects on AK0901 and those on placebo.
Changes in systolic blood pressure during the study | From Baseline to Day 33
  To explore the difference in systolic blood pressure (mmHg) with clinical significance between subjects on AK0901 and those on placebo.
Changes in diastolic blood pressure during the study | From Baseline to Day 33
  To explore the difference in diastolic blood pressure (mmHg) with clinical significance between subjects on AK0901 and those on placebo.
Change from baseline in QT intervals from resting EKGs | Screen/day -1/day1/day14/day28/day33
  EKGs will be performed after the subject has been supine for at least 3 minutes
Change from baseline in QTcF intervals from resting EKGs | Screen/day -1/day1/day14/day28/day33
  EKGs will be performed after the subject has been supine for at least 3 minutes
Change from baseline in heart rate resting EKGs | Screen/day -1/day1/day14/day28/day33
  EKGs will be performed after the subject has been supine for at least 3 minutes
Change from baseline in QRS intervals from resting EKGs | Screen/day -1/day1/day14/day28/day33
  EKGs will be performed after the subject has been supine for at least 3 minutes
Change from baseline in PR intervals from resting EKGs | Screen/day -1/day1/day14/day28/day33
  EKGs will be performed after the subject has been supine for at least 3 minutes
Change in CSHQ score from baseline to each visit in the Double-Blind Treatment Period | From Baseline to Day 33
  Children's Sleep Habits Questionnaire is a retrospective questionnaire containing 33 entries to examine sleep behavior in children. Entries in the key sleep domain are scored on a 3-point scale.A decreasing value of the total score represents a clinical improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing Hu, Study Chair — Clinical Operation Head; Jun Qi, Study Director — Medicial Director
Locations (2):
- China (2):
  - Beijing anding hospital capital medical university, Beijing, Beijing Municipality
  - Peking university sixth hospital, Beijing, Beijing Municipality